CLINICAL TRIAL: NCT01849393
Title: Incentives and Technology Survey 2013: Evaluation of Acceptance of Incentive-Based Adherence Programs and Electronic Medication Monitoring Among HIV-Positive Adolescents
Brief Title: Evaluating Rewards-Based Adherence and Electronic Medication Monitoring in HIV-Positive Adolescents
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: INTECH
Record Dates: First submitted 2013-05-06; First posted 2013-05-08 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-12

CONDITIONS: Human Immunodeficiency Virus (HIV); Acquired Immunodeficiency Syndrome (AIDS)
Keywords: Adolescents; Medication Compliance; Rewards-Based Incentive Programs
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Medication Adherence | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study Population: Participants must meet the eligibility requirements will complete a questionnaire on the computer.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Participants who consent to participate in this study will complete a short questionnaire. The survey will be completely anonymous (not matched with the participant's name). Estimated time to complete the survey is 10-20 minutes.
  Other Names: Survey

SUMMARY:
The primary objective of this project is to assess the study population's acceptance of two medication adherence support strategies: incentive-based programs and electronic medication monitoring. The study population is adolescents (ages 16 - 24) positive for human immunodeficiency virus (HIV) currently undergoing treatment with antiretrovirals at St. Jude's HIV clinic. Participation in the study will involve completion of a survey: an Audio Computer Assisted Self Interview (ACASI). The duration of the survey is anticipated to be 10-20 minutes. Patient identifiers will not be attached the survey.

DETAILED DESCRIPTION:
Whether or not patients take their medications is one of the most noticeable and important predictors of treatment success or failure for HIV infection. Ways to improve compliance, specifically rewards-based programs and electronic medication monitoring, have shown some success in limited clinical research studies focused on adult subjects. Because the social and developmental factors in adolescents are different from adults, adolescents may not respond to these interventions in the same way as adults. This study will investigate adolescent acceptance and the effectiveness of these programs.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive
* Ages 16-24 years.
* Participants must understand written or spoken English, because the ACASI used in the study can only be administered in English.

Exclusion Criteria:

* Adolescents with a documented diagnosis of mental retardation or a significant motor or sensory impairment that would preclude participation in the study survey.

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: HIV-positive adolescents between the ages of 16 and 24 years who are currently undergoing treatment with antiretrovirals at St. Jude's HIV clinic.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Reported perceptions about incentive-based adherence programs and electronic medication monitoring | Once, at enrollment
  Participants will complete a survey/questionnaire on the computer describing their disease state, the frequency and amount of medication taken daily, and how well they comply with taking their medications and attending their clinic appointments. They will also note their perceptions about how incentive-based adherence programs and electronic medication monitoring. Descriptive statistics will be prepared from survey results.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Westfall, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org